CLINICAL TRIAL: NCT04648631
Title: The Microbiome of Hidradenitis Suppurativa (HS) Tunneling Wounds
Brief Title: Hidradenitis Suppurativa (HS) Tunneling Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Next Science LLC (Unknown)
Responsible Party: Principal Investigator, Hadar Lev-Tov, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20201035
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Hidradenitis Suppurativa
Keywords: tunneling wound
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ABWG (Experimental): The participants in this group will be receiving the ABWG daily for 4 consecutive weeks.
  Interventions: Device: antibiofilm surfactant wound gel (ABWG)

INTERVENTIONS:
Device: antibiofilm surfactant wound gel (ABWG) — ABWG is a hydro-gel applied topically using a tongue depressor

SUMMARY:
The purpose of this study is to look at the change in the microbiome (bacterial composition) of an HS tunneling wound and examine if treatment with an antibiofilm surfactant wound gel (ABWG) (a topical medication that will fight bacteria attached to the surface of those tunnels) changes the bacterial composition of the wounds.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years old and older
2. Have diagnosis of HS confirmed by a dermatologist
3. Have at least one HS related tunneling wound that is at least 2 centimeters in length
4. Able to provide informed consent

Exclusion Criteria:

1. Individuals who are not yet adults
2. Women known to be pregnant
3. Prisoners
4. Subjects, who in the opinion of the PI, cannot comply with home application of the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Lev-Tov, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Antibiofilm Surfactant Wound Gel (ABWG): The participants in this group will be receiving the ABWG daily for 4 consecutive weeks. Antibiofilm surfactant wound gel (ABWG): ABWG is a hydro-gel that will be applied topically to both punch sites using a tongue depressor. In the days between visits, patients will apply one fingertip unit of the ABWG to the study wound daily.
Period: Overall Study
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Microbiome
Description: As measured by quantitative 16s rDNA Polymerase Chain Reaction for bacterial enumeration from punch biopsy samples.
Time Frame: Baseline, 4 weeks
Population: Only 8 patients of the 15 had with enough tissue sample for analysis.
Measure: Mean (Standard Deviation); unit: colony forming units per ml (CFU/ml)
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
Number analyzed (Participants) | 8
colony forming units per ml (CFU/ml)
  Baseline | 5.46 (1.85)
  4 weeks | 3.88 (1.09)

2. Secondary Outcome: Change in Lesion Severity as Measured by HS-PGA
Description: HS Physician's Global Assessment (HS-PGA) Scale is a 6 point Likert scale from 0 (clear) to 5 (very severe)
Time Frame: Baseline, 4 week
Population: this was an oversight of the translation of the protocol to the CRF that resulted in the 4 week data point not collected.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
Number analyzed (Participants) | 15
units on a scale
  Baseline | 3.00 [2.00 to 5.00]
  4 weeks: number analyzed (Participants) | 0

3. Secondary Outcome: Change in Lesion Severity as Measured by the Hurley Stage
Description: The Hurley score is staged as: 1 (single or multiple abscesses without sinus tract formation or scarring); 2 (recurrent abscesses with one or more sinus tracts and scarring widely separated by normal skin); 3 (diffuse involvement with multiple sinus tracts and no intervening normal skin).
Time Frame: Baseline, 4 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
Number analyzed (Participants) | 15
score on a scale
  Baseline | 2.00 [2.00 to 3.00]
  4 weeks: number analyzed (Participants) | 0

4. Secondary Outcome: Change in Pain as Measured by VAS
Description: Visual Analog Scale (VAS) has a total score ranging from 0 to 10 with the higher score indicating greater pain.
Time Frame: Baseline, 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
Number analyzed (Participants) | 15
units on a scale
  Baseline | 1.40 [0.34 to 2.64]
  4 weeks | 0.96 [0.05 to 3.56]

5. Secondary Outcome: Change HS Lesion Erythema
Description: As measured the Clinician Erythema Assessment (CEA) scale. CEA scale ranges from 0 (clear) to 4 (severe).
Time Frame: Baseline, 4 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
Number analyzed (Participants) | 15
score on a scale
  Baseline | 1.00 [0.00 to 3.00]
  4 weeks | 2.00 [0.00 to 3.00]

6. Secondary Outcome: Change in Exudate
Description: Exudate will be evaluated using a 5 point Likert scale from 0 (Dry) to 4 (Leaking).
Time Frame: Baseline, 4 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
Number analyzed (Participants) | 15
score on a scale
  Baseline | 0.00 [0.00 to 2.00]
  4 weeks | 0.00 [0.00 to 2.00]

7. Secondary Outcome: Change in Range of Motion
Description: As measured by goniometer
Time Frame: Baseline, 4 weeks
Population: Data for this outcome measure was not collected due to instrument needed for outcome measure was never received for the study, impeding the collection of this specific data point at both baseline and "4 weeks" timepoint.
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With Decreased Pain Medication Use
Description: Pain medication use will be reported as the number of participants that reports a decrease in the dose and/or frequency of pain medication use
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
Number analyzed (Participants) | 15
participants | 4

9. Secondary Outcome: Number of Participants With Escalated Pain Medication Use
Description: Pain medication use will be reported as the number of participants that reports an escalation from using Non-steroidal Anti-inflammatory Drugs (NSAIDs)/acetaminophen to opioids
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
Number analyzed (Participants) | 15
participants | 1

10. Secondary Outcome: Change in Number of Days of Work/School Lost
Description: As self-reported by participants the number of days missed over the length of the study.
Time Frame: Baseline, 4 weeks
Measure: Median (Full Range); unit: Days
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
Number analyzed (Participants) | 15
Days
  Baseline | 0.00 [0.00 to 2.00]
  4 weeks | 0.00 [0.00 to 3.00]

11. Secondary Outcome: Number of Dressings Used
Description: As reported by participants
Time Frame: 4 weeks
Measure: Median (Full Range); unit: number of dressings
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
Number analyzed (Participants) | 15
number of dressings | 13.00 [0.00 to 20.00]

12. Secondary Outcome: Change in Quality of Life as Measured by HiSQOL
Description: HS quality of life (HiSQOL) has a total score ranging from 0 to 68, with higher scores indicating more severe impact on participant's quality of life
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
Number analyzed (Participants) | 15
score on a scale
  Baseline | 44.00 (14.04)
  4 weeks | 44.80 (20.41)

13. Secondary Outcome: Change in Quality of Life as Measured by DLQI
Description: Dermatology Life Quality Index (DLQI) has a total score ranging from 0 to 30 with the lower score indicating higher health related quality of life
Time Frame: Baseline, 4 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
Number analyzed (Participants) | 15
score on a scale
  Baseline | 12.00 [2.00 to 30.00]
  4 weeks | 8.00 [0.00 to 25.00]

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Antibiofilm Surfactant Wound Gel (ABWG): The participants in this group will be receiving the ABWG daily for 4 consecutive weeks.
  antibiofilm surfactant wound gel (ABWG): ABWG is a hydro-gel applied topically using a tongue depressor
Arm/Group | Antibiofilm Surfactant Wound Gel (ABWG)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 6/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antibiofilm Surfactant Wound Gel (ABWG) (N=15)
Stinging (Skin and subcutaneous tissue disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT04648631/Prot_000.pdf